CLINICAL TRIAL: NCT05369273
Title: Addition of Platelet Rich Plasma (PRP) in Microfat Lipofilling (MG) in the Treatment of Cranial Flap Scars: A Randomized, Double-blind, Superiority Study
Acronym: LIPOPREP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-A02972-37
Record Dates: First submitted 2022-03-16; First posted 2022-05-11 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Facial Lipofilling
MeSH Terms: interventions — Injections, Intra-Articular

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- adipose graft + Platelet Rich Plasma (Experimental)
  Interventions: Other: intra-articular injection; Radiation: RMI SCANS; Other: RMI SCANS; Other: RMI SCAN
- adipose graft (Other)
  Interventions: Other: intra-articular injection; Radiation: RMI SCANS; Other: RMI SCANS; Other: RMI SCAN

INTERVENTIONS:
Other: intra-articular injection — intra-articular injection
Radiation: RMI SCANS — AT 1 MONTHS BEFORE THE INTERVENTION
Other: RMI SCANS — AT 1MONTH AFTER THE INTERVENTION
Other: RMI SCAN — AT 6 MONTHS AFTER THE INTERVENTION

SUMMARY:
The objective is to show the superiority of the PRP + microfat (MG) mixture compared to microfat alone, in the filling of large subcutaneous depressions of the face and skull. The investigators chose to study the post neurosurgical sequelae after removal and reinstallation of the cranial flap, with, for example, damage to the temporal muscle and asymmetry of the temples or sinking of the cranial flap

DETAILED DESCRIPTION:
This clinical superiority study will be conducted in a double-blind, randomized fashion. The follow-up of each patient will be 6 months post injection.

22 patients will be included and randomized into 2 arms: PRP + microfat or microfat alone. The primary endpoint will be assessed by a radiologist in a blinded fashion, using 3 MRI scans: the month before the procedure, the day after, and at 6 months (time at which fat resorption decreases).

ELIGIBILITY:
Inclusion Criteria:

* Men and women of age
* Desiring a procedure with an aesthetic aim
* Having a minimum of 6 months after the neurosurgical procedure for cranial flap replacement
* In the absence of need for neurosurgical revision,
* Informed consent signed by the patient
* Be affiliated with the health insurance

Exclusion Criteria:

* Contraindication to MRI
* Patients who have already undergone lipofilling at the site of interest before inclusion in the study.
* Contraindication to general anesthesia
* Considered neurosurgical revision
* Carcinological neurosurgery (With the exception of benign tumors with complete excision and/or non-evolving residue requiring no further treatment)
* Healing of the site of interest not acquired at the 1st consultation
* BMI > 35
* Thrombocytopenia< 150 G/L
* Thrombocytosis > 450 G/L
* Known thrombopathy
* HB anemia < 10g/dl
* Active HIV1 and 2 infections, Agp24, HCV Ac, HbS Ag and AcHbc, HTLV I and II Ac, TPHA
* Chronic treatment with corticoids or NSAIDs or anticoagulant
* Immune deficiency
* Infectious diseases
* Minors
* Pregnant or breastfeeding women
* Patient participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
resorption rate of the injected fat | 6 months
  calculated from volumetric measurements assessed from MRI 2 (post-injection) and MRI3 (at 6 months): V MRI 2 - V MRI3

SECONDARY OUTCOMES:
Visual Analogical Pain Scale | 6 MONTHS
  The measurement of the impact of pain on the cranial scar will be evaluated using a visual analog scale (VAS), rated from 0 to 100.
SF-36 Quality of Life Questionnaire | 6MONTHS
  The Short Form (36) Health Survey is a standardized test for measuring quality of life. It is a measure of health status.
  A score for each dimension of the SF-36 was calculated, ranging from 0 to 100

CONTACTS AND LOCATIONS:
Overall Officials: FRANCOIS CREMIEUX, Study Director — ASSISTANCE PUBLIQUE HOPITAUX MARSEILLE
Locations (1):
- Assiatnce Publique Hopitaux de Marseille, Marseille, Bouche DU Rhone, France